CLINICAL TRIAL: NCT07078006
Title: Efficacy of Injectable Platelet Rich Fibrin Versus Platelet Rich Plasma Injection in Degenerative Temporomandibular Joint
Brief Title: Injectable Platelet Rich Fibrin Versus Platelet Rich Plasma Injection in Degenerative Temporomandibular Joint
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nasser Institute For Research and Treatment (Other Government)
Responsible Party: Principal Investigator, Omar Samir, Oral and Maxillofacial Surgery Department, Faculty of Oral & Dental Medicine, AL Azhar University, Assuit, Egypt., Nasser Institute For Research and Treatment
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 55653465
Record Dates: First submitted 2024-12-31; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Platelet Rich Fibrin; Platelet Rich Plasma Injection; Degenerative Temporomandibular Joint

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Group I (Experimental): Patients underwent arthrocentesis followed by a platelet-rich fibrin (PRF) injection using a conventional temporomandibular joint (TMJ) injection technique, aided by facial anatomical landmarks.
  Interventions: Other: Platelet Rich Fibrin
- Group II (Active Comparator): Patients underwent arthrocentesis followed by a platelet-rich plasma (PRP) injection using a conventional temporomandibular joint (TMJ) injection technique, aided by facial anatomical landmarks.
  Interventions: Other: Platelet Rich Plasma

INTERVENTIONS:
Other: Platelet Rich Fibrin — Patients underwent arthrocentesis followed by a platelet-rich fibrin (PRF) injection using a conventional temporomandibular joint (TMJ) injection technique, aided by facial anatomical landmarks.
  Arms: Group I
Other: Platelet Rich Plasma — Patients underwent arthrocentesis followed by a platelet-rich plasma (PRP) injection using a conventional temporomandibular joint (TMJ) injection technique, aided by facial anatomical landmarks.
  Arms: Group II

SUMMARY:
The study aimed to compare the efficacy of injectable platelet rich fibrin (I-PRF) versus platelet rich plasma (PRP) injection in degenerative temporomandibular joint (TMJ).

DETAILED DESCRIPTION:
Degenerative joint disease (DJD), a frequently observed as osteoarthritic condition in clinical practice, manifests as a persistent and continuous transformation in joint configuration due to the deterioration and attrition of articular cartilage, accompanied by modifications in the subchondral bone and other soft tissue.

Treatment includes physical therapy, pulsed electrical stimulation, pharmacological, topical ointments, supplements, steroid injections, hyaluronic acid (HA) injections, and acupuncture.

Further studies have been carried out to better investigate the effectiveness of different techniques to perform arthrocentesis by using growth factors, autologous solutions, or alternative materials; the materials most used are platelet-rich plasma (PRP) and HA in arthrocentesis or by injection.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years old.
* Both sexes.
* Patients with unilateral or bilateral temporomandibular joint (TMJ) osteoarthritis according to magnetic resonance imaging (MRI) evaluation.

Exclusion Criteria:

* Patients under any type of antiplatelet or anticoagulant medications.
* Cardiovascular, renal, or hepatic disease.
* Diabetes.
* Anemia.
* Vascular insufficiency.
* Peripheral neuropathy.
* Previous surgery for TMJ and rheumatoid arthritis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2024-07-23 (Actual)

PRIMARY OUTCOMES:
Pain improvement | 6 months post-procedure
  Each patient will be instructed about postoperative pain assessment with the Visual Analogue Scale (VAS). VAS (0 represents "no pain" while 10 represents "the worst pain imaginable"). VAS was recorded preoperatively, immediately after the procedures, 1 month, 3 months, and 6 months postoperatively.

SECONDARY OUTCOMES:
Assessment of tissue repair | 6 months post-procedure
  Tissue repair in the form of initiating fibrin coating around the osteoarthritic joint by using Magnetic Resonance Imaging (MRI) was recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Nasser, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.